CLINICAL TRIAL: NCT04909112
Title: Olfactory and Taste Disturbances in Sjogren's Syndrome
Acronym: TOG_SJOGREN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-007-TOG_SJOGREN
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Sjogren's Syndrome
Keywords: Sjogren's syndrome; olfactory disorder; taste disorder; (intra-nasal and oral) trigeminal impairments
MeSH Terms: conditions — Sjogren's Syndrome; Taste Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1: patients with Sjogren's syndrome (Other): Patients with Sjogren's syndrome
  Interventions: Other: Evaluation of olfactory function; Other: Evaluation of taste function; Other: Evaluation of (intra-nasal and oral) trigeminal functions
- group 2: patients without sicca syndrome (Other): Patients without sicca syndrome
  Interventions: Other: Evaluation of olfactory function; Other: Evaluation of taste function; Other: Evaluation of (intra-nasal and oral) trigeminal functions

INTERVENTIONS:
Other: Evaluation of olfactory function — Evaluation of olfactory function using olfactory detection thresholds
Other: Evaluation of taste function — Evaluation of taste function using taste detection thresholds
Other: Evaluation of (intra-nasal and oral) trigeminal functions — Evaluation of (intra-nasal and oral) trigeminal, interacting with olfactory and taste pathways, using odor and taste stimuli.

SUMMARY:
Sjögren syndrome is an autoimmune disease, responsible for xerostomia and xerophthalmia. Other organs and tissues can be affected: the skin, vaginal and nasal mucous membranes. As well, olfactory disorders have been also described in Sjögren syndrome.

Xerostomia often causes significant functional impairment of taste function. Impairment of taste function has been poorly evaluated in Sjögren syndrome like olfactory or (intra-nasal and oral) trigeminal disorders.

DETAILED DESCRIPTION:
The aim of the study is to evaluate olfactory, taste (intra-nasal and oral) trigeminal functions in patients with Sjogren's syndrome compared to patients without sicca syndrome.

ELIGIBILITY:
Inclusion Criteria:

* group 1 : patients with Sjogren's syndrome
* group 2: patients without sicca syndrome
* older than 18 years old
* consenting to participate to the study

Exclusion Criteria:

* smoking patients
* patients with stomatitis
* patients with upper respiratory tract infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Olfactory detection thresholds for Phenyl-ethyl alcohol | Day 0
  Successive dilutions of odorants by a factor 2 will be realized with distilled water as solvent.
  The odorant stimulus will be presented in a white glass bottle filled with 4 ml of liquid. The bottle will be presented for 3 seconds, medially 1 cm under both nostrils. Odour thresholds will be assessed using an ascending staircase, binary (stimulus vs. blank) forced-choice procedure, with inter-trial intervals of 90 seconds. The two bottles will presented to the subject in random order. After sniffing each stimulus, the participant will be asked to identify the one who smelled stronger. An incorrect choice will led to increase the concentration of the stimulus in the next trial. The dilution step at which the odorant stimulus will be first detected correctly three times in a row will be recorded as the detection threshold.
Olfactory detection thresholds for Butanol | Day 0
  Successive dilutions of odorants by a factor 2 will be realized with distilled water as solvent.
  The odorant stimulus will be presented in a white glass bottle filled with 4 ml of liquid. The bottle will be presented for 3 seconds, medially 1 cm under both nostrils. Odour thresholds will be assessed using an ascending staircase, binary (stimulus vs. blank) forced-choice procedure, with inter-trial intervals of 90 seconds. The two bottles will presented to the subject in random order. After sniffing each stimulus, the participant will be asked to identify the one who smelled stronger. An incorrect choice will led to increase the concentration of the stimulus in the next trial. The dilution step at which the odorant stimulus will be first detected correctly three times in a row will be recorded as the detection threshold.
Olfactory detection thresholds for Pyridine | Day 0
  Successive dilutions of odorants by a factor 2 will be realized with distilled water as solvent.
  The odorant stimulus will be presented in a white glass bottle filled with 4 ml of liquid. The bottle will be presented for 3 seconds, medially 1 cm under both nostrils. Odour thresholds will be assessed using an ascending staircase, binary (stimulus vs. blank) forced-choice procedure, with inter-trial intervals of 90 seconds. The two bottles will presented to the subject in random order. After sniffing each stimulus, the participant will be asked to identify the one who smelled stronger. An incorrect choice will led to increase the concentration of the stimulus in the next trial. The dilution step at which the odorant stimulus will be first detected correctly three times in a row will be recorded as the detection threshold.

SECONDARY OUTCOMES:
Taste detection thresholds for salty taste | Day 0
  Taste strips will be placed on the tongue. Each strip contains a stimulus at different concentrations. Patient will be asked if he/she perceive the taste.
Taste detection thresholds for sweet taste | Day 0
  Taste strips will be placed on the tongue. Each strip contains a stimulus at different concentrations. Patient will be asked if he/she perceive the taste.
Taste detection thresholds for sour taste | Day 0
  Taste strips will be placed on the tongue. Each strip contains a stimulus at different concentrations. Patient will be asked if he/she perceive the taste.
Taste detection thresholds for bitter taste | Day 0
  Taste strips will be placed on the tongue. Each strip contains a stimulus at different concentrations. Patient will be asked if he/she perceive the taste.
Taste detection thresholds for trigeminal stimuli | Day 0
  Taste strips will be placed on the tongue. Each strip contains a stimulus at different concentrations. Patient will be asked if he/she perceive the taste.

CONTACTS AND LOCATIONS:
Overall Officials: Clovis FOGUEM, MD, Principal Investigator — Université de Reims Champagne-Ardenne
Locations (1):
- Université de Reims Champagne-Ardenne, Reims, France